CLINICAL TRIAL: NCT01177059
Title: A Long Term Follow-up Protocol to Evaluate the Safety and Survival of Autologous CD34+ Hematopoietic Progenitor Cells Transduced With an Anti-HIV-1 Ribozyme (OZ1) in Patients With HIV-1 Infection
Brief Title: Long Term Follow-Up Study of Human Immunodeficiency Virus Type 1 (HIV-1) Positive Patients Who Have Received OZ1 Gene Therapy as Part of a Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR016027; OZ1-HV1-202 (Other: Janssen-Cilag Pty Ltd, Australia)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: HIV-1
Keywords: Gene Therapy; Anti-HIV-1 Ribozyme; OZ1; HIV-1 Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Anti-HIV-1 Ribozyme (OZ1) transduced cells (Other): OZ1 transduced cells Long term follow up of previously infused OZ1 transduced cells
  Interventions: Genetic: OZ1 transduced cells

INTERVENTIONS:
Genetic: OZ1 transduced cells — Long term follow up of previously infused OZ1 transduced cells

SUMMARY:
The purpose of this Observational Study is long term follow-up of the Human Immunodeficiency Virus -1 (HIV-1) infected patients who have received a gene therapy product (anti-HIV-1 Ribozyme [OZ1]) as part of an earlier phase 2 trial. Patients are seen twice yearly until 5 years from initial infusion of study drug has elapsed and then yearly until withdrawal or study completion. The study will monitor for and record any ill effects from the gene therapy product to provide long term safety information.

DETAILED DESCRIPTION:
During an earlier phase 2 base trial (study # NCT00074997), HIV-1 infected patients received a gene therapy product (anti-HIV-1 Ribozyme [OZ1]). Gene therapy is an investigational treatment where genes are inserted into an individual's cells and tissues to treat a disease. The gene therapy OZ1 is thought to have anti-HIV-1 actions. This is an Observational Study to provide long term follow-up of those HIV-1 infected patients who received the gene therapy product (anti-HIV-1 Ribozyme [OZ1]) as part of the earlier study. Patients are seen twice yearly until 5 years from initial infusion of study drug has elapsed and then yearly until withdrawal or study completion. The study will monitor for and record any ill effects from the gene therapy product to provide long term safety information. Observational study - no investigational drug administered.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were enrolled (between 18 and 45 years of age) in the base study "OTH/OZ1-INT-1" (NCT00074997) will be invited to participate in this long term follow-up study
* Patients must have received the Final Cell Product infusion in base study "OTH/OZ1-INT-1"
* Have signed Informed Consent Form

Exclusion Criteria:

* All patients who were enrolled in the OTH/OZ1-INT-1 study and received the final cell product will be invited to participate in this long term follow-up study. After unblinding of the OTH/OZ1-INT-1 study, any patients in the placebo arm will be withdrawn from this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-12-06 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (6):
- United States (3):
  - Los Angeles, California
  - San Francisco, California
  - New York, New York
- Australia (3):
  - Darlinghurst
  - Surry Hills
  - Sydney

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed original study (OTH/OZ1-INT-1 [NCT00074997]) were enrolled in this long term follow-up (LTFU) study. After unblinding of original study, participants in placebo group were withdrawn from LTFU study, except first participant who received Moloney murine leukemia virus based retroviral vector (LNL6) transduced CD34+ cells.
Groups:
- Anti-HIV-1 Ribozyme (OZ1) Transduced Cells: Participants who received an infusion of final cell product (that is, a cluster of differentiation [CD]34+ cells with or without gene transfer product) in the original study (OTH/OZ1-INT-1) were followed up in this study.
Period: Overall Study
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
Started | 68
Completed | 18
Not Completed | 50
Not completed — Received placebo in OTH/OZ1-INT-1 study | 30
Not completed — Withdrew consent | 2
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Population: The baseline (safety) population included all participants who were enrolled in the original OTH/OZ1-INT-1 study and continued participation in the long term follow-up OZ1-HV1-202/OZ1HIV2001 study.
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 5
  Asian | 2
  Caucasian | 53
  Hispanic | 6
  Maori/Polynesian | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 32
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clonal Expansion of Cells With a Predominant OZ1 Insertion Site
Description: Percentage of participants with clonal expansion of cells with a predominant OZ1 insertion site was reported. A predominant integration site was defined as an integration site which has a density of at least 50 percent (%) of the total signal detected by polymerase chain reaction (PCR), when the percentage of cells marked by vector was greater than (>)1% of the test cell population.
Time Frame: Approximately up to 15 years
Population: Per protocol (PP) population set included all participants in the safety population who received OZ1 or Moloney murine leukemia virus based retroviral vector (LNL6) transduced final cell product in the original OTH/OZ1-INT-1 study.
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
Number analyzed (Participants) | 37
Percentage of participants | 0

2. Primary Outcome: Percentage of Participants With Insertional Oncogenesis
Description: Percentage of participants with insertional oncogenesis by clonal expansion of cells modified with OZ1/LNL6 were reported.
Time Frame: Approximately up to 15 years
Population: Per protocol population set included all participants in the safety population who received OZ1 or LNL6 transduced final cell product in the original OTH/OZ1-INT-1 study.
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
Number analyzed (Participants) | 37
Percentage of participants | 0

3. Primary Outcome: Number of Participants With Quantitative Marking of Gene Transfer Product in Peripheral Blood Mononuclear Cells (PBMC) Over Time
Description: OZ1 and LNL6 marking analysis were performed by quantitative deoxyribonucleic acid-polymerase chain reaction (DNA-PCR). Number of participants in each of 3 categories for gene detection: Not Detected, Detected (1, 2 and 3 of the 3 triplicates of the sample were detected respectively [1/3 Detected, 2/3 Detected, 3/3 Detected]) and Detected (Quantifiable) were reported for marking of gene transfer product in PBMC.
Time Frame: Up to end of study (Approximately up to 15 years)
Population: PP population set included all participants in safety population who received OZ1/LNL6 transduced final cell product in original OTH/OZ1-INT-1 study. Here 'n' specifies participants analyzed for this endpoint at given time point.
Measure: Number; unit: Participants
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
Number analyzed (Participants) | 37
Participants
  2 years post-infusion: Not Detected | 33
  2 years post-infusion: 1/3 Detected | 4
  2 years post-infusion: 2/3 Detected | 0
  2 years post-infusion: 3/3 Detected | 0
  2 years post-infusion: Detected (Quantifiable) | 0
  2.5 years post-infusion: Not Detected: number analyzed (Participants) | 34
  2.5 years post-infusion: Not Detected | 31
  2.5 years post-infusion: 1/3 Detected: number analyzed (Participants) | 34
  2.5 years post-infusion: 1/3 Detected | 2
  2.5 years post-infusion: 2/3 Detected: number analyzed (Participants) | 34
  2.5 years post-infusion: 2/3 Detected | 1
  2.5 years post-infusion: 3/3 Detected: number analyzed (Participants) | 34
  2.5 years post-infusion: 3/3 Detected | 0
  2.5 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 34
  2.5 years post-infusion: Detected (Quantifiable) | 0
  3 years post-infusion: Not Detected: number analyzed (Participants) | 35
  3 years post-infusion: Not Detected | 31
  3 years post-infusion: 1/3 Detected: number analyzed (Participants) | 35
  3 years post-infusion: 1/3 Detected | 3
  3 years post-infusion: 2/3 Detected: number analyzed (Participants) | 35
  3 years post-infusion: 2/3 Detected | 0
  3 years post-infusion: 3/3 Detected: number analyzed (Participants) | 35
  3 years post-infusion: 3/3 Detected | 1
  3 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 35
  3 years post-infusion: Detected (Quantifiable) | 0
  3.5 years post-infusion: Not Detected: number analyzed (Participants) | 28
  3.5 years post-infusion: Not Detected | 28
  3.5 years post-infusion: 1/3 Detected: number analyzed (Participants) | 28
  3.5 years post-infusion: 1/3 Detected | 0
  3.5 years post-infusion: 2/3 Detected: number analyzed (Participants) | 28
  3.5 years post-infusion: 2/3 Detected | 0
  3.5 years post-infusion: 3/3 Detected: number analyzed (Participants) | 28
  3.5 years post-infusion: 3/3 Detected | 0
  3.5 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 28
  3.5 years post-infusion: Detected (Quantifiable) | 0
  4 years post-infusion: Not Detected: number analyzed (Participants) | 32
  4 years post-infusion: Not Detected | 28
  4 years post-infusion: 1/3 Detected: number analyzed (Participants) | 32
  4 years post-infusion: 1/3 Detected | 4
  4 years post-infusion: 2/3 Detected: number analyzed (Participants) | 32
  4 years post-infusion: 2/3 Detected | 0
  4 years post-infusion: 3/3 Detected: number analyzed (Participants) | 32
  4 years post-infusion: 3/3 Detected | 0
  4 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 32
  4 years post-infusion: Detected (Quantifiable) | 0
  4.5 years post-infusion: Not Detected: number analyzed (Participants) | 25
  4.5 years post-infusion: Not Detected | 19
  4.5 years post-infusion: 1/3 Detected: number analyzed (Participants) | 25
  4.5 years post-infusion: 1/3 Detected | 5
  4.5 years post-infusion: 2/3 Detected: number analyzed (Participants) | 25
  4.5 years post-infusion: 2/3 Detected | 1
  4.5 years post-infusion: 3/3 Detected: number analyzed (Participants) | 25
  4.5 years post-infusion: 3/3 Detected | 0
  4.5 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 25
  4.5 years post-infusion: Detected (Quantifiable) | 0
  5 years post-infusion: Not Detected: number analyzed (Participants) | 27
  5 years post-infusion: Not Detected | 27
  5 years post-infusion: 1/3 Detected: number analyzed (Participants) | 27
  5 years post-infusion: 1/3 Detected | 0
  5 years post-infusion: 2/3 Detected: number analyzed (Participants) | 27
  5 years post-infusion: 2/3 Detected | 0
  5 years post-infusion: 3/3 Detected: number analyzed (Participants) | 27
  5 years post-infusion: 3/3 Detected | 0
  5 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 27
  5 years post-infusion: Detected (Quantifiable) | 0
  6 years post-infusion: Not Detected: number analyzed (Participants) | 20
  6 years post-infusion: Not Detected | 18
  6 years post-infusion: 1/3 Detected: number analyzed (Participants) | 20
  6 years post-infusion: 1/3 Detected | 0
  6 years post-infusion: 2/3 Detected: number analyzed (Participants) | 20
  6 years post-infusion: 2/3 Detected | 1
  6 years post-infusion: 3/3 Detected: number analyzed (Participants) | 20
  6 years post-infusion: 3/3 Detected | 0
  6 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 20
  6 years post-infusion: Detected (Quantifiable) | 1
  7 years post-infusion: Not Detected: number analyzed (Participants) | 10
  7 years post-infusion: Not Detected | 9
  7 years post-infusion: 1/3 Detected: number analyzed (Participants) | 10
  7 years post-infusion: 1/3 Detected | 0
  7 years post-infusion: 2/3 Detected: number analyzed (Participants) | 10
  7 years post-infusion: 2/3 Detected | 0
  7 years post-infusion: 3/3 Detected: number analyzed (Participants) | 10
  7 years post-infusion: 3/3 Detected | 1
  7 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 10
  7 years post-infusion: Detected (Quantifiable) | 0
  8 years post-infusion: Not Detected: number analyzed (Participants) | 9
  8 years post-infusion: Not Detected | 9
  8 years post-infusion: 1/3 Detected: number analyzed (Participants) | 9
  8 years post-infusion: 1/3 Detected | 0
  8 years post-infusion: 2/3 Detected: number analyzed (Participants) | 9
  8 years post-infusion: 2/3 Detected | 0
  8 years post-infusion: 3/3 Detected: number analyzed (Participants) | 9
  8 years post-infusion: 3/3 Detected | 0
  8 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 9
  8 years post-infusion: Detected (Quantifiable) | 0
  9 years post-infusion: Not Detected: number analyzed (Participants) | 7
  9 years post-infusion: Not Detected | 6
  9 years post-infusion: 1/3 Detected: number analyzed (Participants) | 7
  9 years post-infusion: 1/3 Detected | 1
  9 years post-infusion: 2/3 Detected: number analyzed (Participants) | 7
  9 years post-infusion: 2/3 Detected | 0
  9 years post-infusion: 3/3 Detected: number analyzed (Participants) | 7
  9 years post-infusion: 3/3 Detected | 0
  9 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 7
  9 years post-infusion: Detected (Quantifiable) | 0
  10 years post-infusion: Not Detected: number analyzed (Participants) | 10
  10 years post-infusion: Not Detected | 9
  10 years post-infusion: 1/3 Detected: number analyzed (Participants) | 10
  10 years post-infusion: 1/3 Detected | 1
  10 years post-infusion: 2/3 Detected: number analyzed (Participants) | 10
  10 years post-infusion: 2/3 Detected | 0
  10 years post-infusion: 3/3 Detected: number analyzed (Participants) | 10
  10 years post-infusion: 3/3 Detected | 0
  10 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 10
  10 years post-infusion: Detected (Quantifiable) | 0
  11 years post-infusion: Not Detected: number analyzed (Participants) | 8
  11 years post-infusion: Not Detected | 7
  11 years post-infusion: 1/3 Detected: number analyzed (Participants) | 8
  11 years post-infusion: 1/3 Detected | 1
  11 years post-infusion: 2/3 Detected: number analyzed (Participants) | 8
  11 years post-infusion: 2/3 Detected | 0
  11 years post-infusion: 3/3 Detected: number analyzed (Participants) | 8
  11 years post-infusion: 3/3 Detected | 0
  11 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 8
  11 years post-infusion: Detected (Quantifiable) | 0
  12 years post-infusion: Not Detected: number analyzed (Participants) | 7
  12 years post-infusion: Not Detected | 7
  12 years post-infusion: 1/3 Detected: number analyzed (Participants) | 7
  12 years post-infusion: 1/3 Detected | 0
  12 years post-infusion: 2/3 Detected: number analyzed (Participants) | 7
  12 years post-infusion: 2/3 Detected | 0
  12 years post-infusion: 3/3 Detected: number analyzed (Participants) | 7
  12 years post-infusion: 3/3 Detected | 0
  12 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 7
  12 years post-infusion: Detected (Quantifiable) | 0
  13 years post-infusion: Not Detected: number analyzed (Participants) | 3
  13 years post-infusion: Not Detected | 3
  13 years post-infusion: 1/3 Detected: number analyzed (Participants) | 3
  13 years post-infusion: 1/3 Detected | 0
  13 years post-infusion: 2/3 Detected: number analyzed (Participants) | 3
  13 years post-infusion: 2/3 Detected | 0
  13 years post-infusion: 3/3 Detected: number analyzed (Participants) | 3
  13 years post-infusion: 3/3 Detected | 0
  13 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 3
  13 years post-infusion: Detected (Quantifiable) | 0
  14 years post-infusion: Not Detected: number analyzed (Participants) | 1
  14 years post-infusion: Not Detected | 1
  14 years post-infusion: 1/3 Detected: number analyzed (Participants) | 1
  14 years post-infusion: 1/3 Detected | 0
  14 years post-infusion: 2/3 Detected: number analyzed (Participants) | 1
  14 years post-infusion: 2/3 Detected | 0
  14 years post-infusion: 3/3 Detected: number analyzed (Participants) | 1
  14 years post-infusion: 3/3 Detected | 0
  14 years post-infusion: Detected (Quantifiable): number analyzed (Participants) | 1
  14 years post-infusion: Detected (Quantifiable) | 0
  End of study: Not Detected: number analyzed (Participants) | 6
  End of study: Not Detected | 6
  End of study: 1/3 Detected: number analyzed (Participants) | 6
  End of study: 1/3 Detected | 0
  End of study: 2/3 Detected: number analyzed (Participants) | 6
  End of study: 2/3 Detected | 0
  End of study: 3/3 Detected: number analyzed (Participants) | 6
  End of study: 3/3 Detected | 0
  End of study: Detected (Quantifiable): number analyzed (Participants) | 6
  End of study: Detected (Quantifiable) | 0

ADVERSE EVENTS:
Time Frame: Approximately up to 15 years
Description: The safety population included all participants who were enrolled in the original OTH/OZ1-INT-1 study and continued participation in the long term follow-up OZ1-HV1-202/OZ1HIV2001 study.
Arm/Group | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 7/68
Other Adverse Events (participants affected / at risk) | 1/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells (N=68)
Rib Fracture (Injury, poisoning and procedural complications) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testicle Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-HIV-1 Ribozyme (OZ1) Transduced Cells (N=68)
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT01177059/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT01177059/SAP_001.pdf